CLINICAL TRIAL: NCT01975987
Title: Identification of Morphological Characteristics to Predict Successful Intubation With the Bonfils Fiberscope
Brief Title: Characteristics to Predict Successful Intubation With the Bonfils Fiberscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13.182
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Endotracheal Intubation
Keywords: Intubation; Bonfils fiberscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubation with the Bonfils fiberscope (Experimental): * Characteristics of patients will be assessed before induction of general anesthesia
  * Glottic visualization will be evaluated by direct laryngoscopy.
  * The endotracheal tube will be loaded onto the scope
  * Intubation will be performed with the Bonfils fiberscope with the patient in supine position with head and neck in neutral position
  * Bonfils fiberscope will be inserted from the right side of the patient's mouth, alongside the molars and advanced underneath the epiglottis. With the tip of the Bonfils in satisfactory position, the endotracheal tube will be advanced into the trachea using gentle rotary motions. The scope will then be removed.
  * Accurate positioning of the endotracheal tube will be confirmed by capnography and lung auscultation.
  Interventions: Device: Bonfils fiberscope

INTERVENTIONS:
Device: Bonfils fiberscope

SUMMARY:
This study is designed to identify patients' features predictive of successful intubation using the Bonfils fiberscope.

Our hypothesis is that some patients' characteristics are predictors of successful intubation with the Bonfils fiberscope.

DETAILED DESCRIPTION:
Endotracheal intubation is an important act in the practice of anesthesiology. Direct laryngoscopy is the most commonly used technique to accomplish this task. Airway characteristics predicting difficult intubation with direct laryngoscopy are well defined. Physical findings, such as Mallampati classification or measurements of the thyromental distance, mouth opening, and neck extension have been validated to help anticipate difficult situations. When direct laryngoscopy is strenuous, early conversion to an alternative technique might reduce the risk of airway compromise and associated morbidity.

Many intubation devices are now available and part of the anesthesiologist's task is to select the alternative approach best suited to each patient's specific features. Despite its use for both elective and unexpectedly difficult intubation, predictive criteria for successful airway management with the Bonfils fiberscope have not been proposed.

The purpose of this study is to identify patients' features, if any, that could predict successful intubation when using the Bonfils fiberscope for perioperative orotracheal intubation in an elective surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients undergoing elective surgery under general anesthesia, requiring endotracheal intubation

Exclusion Criteria:

* Induction planned without neuromuscular blocking agents
* Need for a rapid sequence induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Morphologic and morphometric predictors of successful tracheal intubation with the Bonfils fiberscope | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
  This study will correlate patients' morphometric and morphologic characteristics with the number of attempts and time needed for intubation using the Bonfils fiberscope.

SECONDARY OUTCOMES:
Time to successful intubation | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
Number of attempts to successful intubation | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
Score on the Intubation Difficulty Scale | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
  To calculate the Intubation Difficulty Score the following variables will be collected: number of attempts, number of operators, necessity to use an alternative intubation technique, glottic visualization and effort needed to obtain optimal view of the glottis, necessity of external laryngeal pressure and vocal cords position during intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Robitaille, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada